CLINICAL TRIAL: NCT00887965
Title: A Transiliac Crest Bone Histology and Histomorphometry Study in Postmenopausal Women With Low Bone Mass or Osteoporosis Previously Treated With Denosumab
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 20080287
Record Dates: First submitted 2009-04-23; First posted 2009-04-24 (Estimated); Results first posted 2013-10-17 (Estimated); Last update posted 2013-11-15 (Estimated); Status verified 2013-10

CONDITIONS: Low Bone Mass; Low Bone Mineral Density; Osteoporosis; Postmenopausal Osteoporosis
Keywords: Low Bone Mass; Low Bone Mineral Density; Osteoporosis; Postmenopausal Osteoporosis; Bone Biopsy; Transiliac Crest Bone Histology; Histomorphometry
MeSH Terms: conditions — Bone Diseases, Metabolic; Osteoporosis; Osteoporosis, Postmenopausal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Previous denosumab (Other): Participants who had previously received denosumab received a transiliac crest bone biopsy performed following standard labeling procedures with tetracycline or tetracycline derivative.
  Interventions: Drug: Previous denosumab

INTERVENTIONS:
Drug: Previous denosumab — Participants who had previously received denosumab received a transiliac crest bone biopsy performed following standard labeling procedures with tetracycline or tetracycline derivative.

SUMMARY:
To characterize the effects of discontinuation of denosumab therapy on variables of bone histology in postmenopausal women with low bone mass or osteoporosis. Patients who have received denosumab and completed study 20050179 (NCT00293813), completed study 20050141 (NCT00330460), completed study 20060237 (NCT00515463), completed study 20030216 (NCT00089791) but did not enroll in study 20060289 (NCT00523341) will be included in this study. Patients who will participate in the off-treatment imaging study for 20080747 (NCT00890981) are also eligible.

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory postmenopausal women
* Received denosumab and completed study 20050179 (NCT00293813), completed study 20050141 (NCT00330460), completed study 20060237 (NCT00515463), completed study 20030216 (NCT00089791) but did not enroll in study 20060289 (NCT00523341). Patients who will participate in the off-treatment imaging study for 20080747 (NCT00890981) also are eligible.
* Completed participation in eligible studies ≥ 12 and ≤ 36 months prior to screening
* Provide signed informed consent

Exclusion Criteria:

* Did not receive denosumab in studies 20050141, 20060237, 20030216, or 20050179.
* Discontinued investigational product before end of study visit for studies 20050141, 20060237, 20030216, or 20050179.
* Received > 1 month osteoporosis treatment since having completed studies 20050141, 20060237, 20030216, or 20050179.
* Received zoledronic acid at any time after ending study participation in parent studies 20050141, 20050179, 20030216, or 20060237.
* Newly diagnosed with any of the following conditions during the intervening period since completing studies 20050141, 20060237, 20030216, or 20050179:
* Hyperthyroidism (stable on anti-thyroid therapy or post-ablation is allowed, if the Thyroid Stimulating Hormone is within the normal range)
* Hypothyroidism (stable on thyroid replacement therapy is allowed, if the Thyroid Stimulating Hormone is within the normal range)
* Hyper- or hypoparathyroidism
* Osteomalacia
* Paget's disease of bone
* Other bone diseases which affect bone metabolism (eg, osteopetrosis, osteogenesis imperfecta)
* Malignancy within the last 5 years (except cervical carcinoma in situ or basal cell carcinoma).
* Self-reported alcohol or drug abuse within the previous 12 months.
* Permanently non-ambulatory subjects (use of assistive device eg cane, walker is permitted).
* Has known or suspected sensitivity or contraindication to tetracycline derivatives.
* Received any investigational product other than denosumab.
* Current use of the following osteoporosis agents: bisphosphonates, calcitonin, fluoride, parathyroid hormone analogue, selective estrogen receptor modulators, systemic oral or transdermal estrogen (except vaginal preparations and estrogen creams which are acceptable), strontium or tibolone.
* Has undergone bilateral transiliac crest bone biopsy in the past.
* Current use of medications that, in the opinion of the investigator, cannot be discontinued and may compromise the safety of the subject when undergoing the bone biopsy procedure (eg, aspirin, warfarin, high-dose heparin).
* Current use of systemic glucocorticoid therapy (topical or nasal steroids are permitted).
* Evidence of coagulopathy that in the opinion of the investigator, may compromise patient safety when subjected to the bone biopsy procedure.
* Any disorder that, in the opinion of the investigator, may compromise the ability of the participant to give written informed consent and/or comply with study procedures.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2009-06; Primary Completion 2010-06 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First subject enrolled on 02-JUN-09. Last subject enrolled on 28-APR-2010.
Groups:
- Previous Denosumab: Participants who had previously received Denosumab 60 mg every 6 months and had transiliac bone biopsy.
Period: Overall Study
Arm/Group | Previous Denosumab
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Previous Denosumab
Number analyzed (Participants) | 15
Age Continuous [Mean (Standard Deviation); unit: Years] | 62.1 (5.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 0
Ethnic group: White or Caucasian [Number; unit: Participants] | 15

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Normal/Abnormal Bone Histology
Description: The number of participants with normal/abnormal bone histology as assessed by bone biopsy samples at the central histomorphometric facility. Normal bone histology is characterized by: - normal lamellar bone, - normal mineralization or - osteoid (the organic matrix of bone; young bone that has not undergone calcification). Biopsies with abnormal bone histology are characterized by: - osteomalacia, - marrow fibrosis, - clinically significant marrow abnormality or - woven bone.
Time Frame: 25-34 days post-Day 1
Population: All enrolled patients who had at least one evaluable biopsy
Measure: Number; unit: Participants
Arm/Group | Previous Denosumab
Number analyzed (Participants) | 15
Participants
  Normal lamellar bone | 15
  Normal mineralization | 15
  Osteoid | 15
  Osteomalacia | 0
  Marrow fibrosis | 0
  Clinically significant marrow abnormality | 0
  Woven bone | 0

2. Secondary Outcome: Bone Histomorphometry: Cancellous Bone Volume
Description: Cancellous (trabecular) bone volume (Tb.V) is the relative volume of total cancellous bone measured (TV), expressed as percentage, that is occupied by trabeculae. Cancellous bone volume was measured using Fluorochrome labeling with tetracyclene and tartrate-resistant acid phosphatase stain (TRAP) staining techniques.
Time Frame: 25-34 days post-Day 1
Population: All enrolled patients with at least one biopsy evaluable for histomorphometry
Measure: Median (Inter-Quartile Range); unit: percentage of total volume
Arm/Group | Previous Denosumab
Number analyzed (Participants) | 14
percentage of total volume
  Fluorochrome labeling | 13.765 [10.190 to 18.080]
  TRAP staining | 17.320 [12.540 to 23.230]

3. Secondary Outcome: Bone Histomorphometry: Trabecular Number
Description: Trabecular number (Tb.N) is the number of trabeculae present per lineal mm and is calculated as trabecular bone volume/trabecular thickness. Tb.N is a measure of trabecular connectivity and decreases with bone loss.
Time Frame: 25-34 days post-Day 1
Population: All enrolled patients with at least one biopsy evaluable for histomorphometry.
Measure: Median (Inter-Quartile Range); unit: mm^-1
Arm/Group | Previous Denosumab
Number analyzed (Participants) | 14
mm^-1 | 1.050 [1.000 to 1.160]

4. Secondary Outcome: Bone Histomorphometry: Trabecular Separation
Description: Trabecular separation (Tb.Sp) is the mean distance in mm between trabeculae (measured by integrated computer graphics). Tb.Sp increases with trabecular bone loss.
Time Frame: 25-34 days post-Day 1
Population: All enrolled patients with at least one biopsy evaluable for histomorphometry.
Measure: Median (Inter-Quartile Range); unit: μm
Arm/Group | Previous Denosumab
Number analyzed (Participants) | 14
μm | 807.270 [705.690 to 896.110]

5. Secondary Outcome: Bone Histomorphometry: Trabecular Thickness
Description: Mean trabecular thickness (Tb.Th) is a measure of trabecular structure and is calculated as the reciprocal of total bone (trabecular) surfaces. Tb.Th is reduced by aging and osteoporosis.
Time Frame: 25-34 days post-Day 1
Population: All enrolled patients with at least one biopsy evaluable for histomorphometry.
Measure: Median (Inter-Quartile Range); unit: μm
Arm/Group | Previous Denosumab
Number analyzed (Participants) | 14
μm | 131.465 [117.090 to 159.030]

6. Secondary Outcome: Bone Histomorphometry: Cortical Width
Description: Cortical width correlates with dual photon absorptiometric (DPX) measurements of bone density.
Time Frame: 25-34 days post-Day 1
Population: All enrolled patients with at least one biopsy evaluable for histomorphometry.
Measure: Median (Inter-Quartile Range); unit: μm
Arm/Group | Previous Denosumab
Number analyzed (Participants) | 14
μm | 747.45 [524.50 to 845.40]

7. Secondary Outcome: Bone Histomorphometry: Surface Density
Description: Surface density is calculated by total bone (trabecular) surfaces / total tissue volume.
Time Frame: 25-34 days post-Day 1
Population: All enrolled patients with at least one biopsy evaluable for histomorphometry.
Measure: Median (Inter-Quartile Range); unit: mm^2 /mm^3
Arm/Group | Previous Denosumab
Number analyzed (Participants) | 14
mm^2 /mm^3 | 2.110 [2.000 to 2.320]

8. Secondary Outcome: Bone Histomorphometry: Osteoblast - Osteoid Interface
Description: Osteoblast - osteoid interface is calculated as osteoblast surface / osteoid surface * 100.
Time Frame: 25-34 days post-Day 1
Population: All enrolled patients with at least one biopsy evaluable for histomorphometry.
Measure: Median (Inter-Quartile Range); unit: percentage of osteoid surface
Arm/Group | Previous Denosumab
Number analyzed (Participants) | 14
percentage of osteoid surface | 30.165 [8.990 to 41.210]

9. Secondary Outcome: Bone Histomorphometry: Osteoid Surface
Description: Osteoid surface is expressed as a percentage total bone surface.
Time Frame: 25-34 days post-Day 1
Population: All enrolled patients with at least one biopsy evaluable for histomorphometry.
Measure: Median (Inter-Quartile Range); unit: percentage of bone surface
Arm/Group | Previous Denosumab
Number analyzed (Participants) | 14
percentage of bone surface | 3.280 [1.200 to 8.370]

10. Secondary Outcome: Bone Histomorphometry: Osteoid Width
Description: Osteoid thickness (width; O.Th) is the mean thickness of osteoid seams on cancellous surfaces. O.Th is normally <12.5 µm. Increased O.Th suggests abnormal mineralization (osteomalacia).
Time Frame: 25-34 days post-Day 1
Population: All enrolled patients with at least one biopsy evaluable for histomorphometry.
Measure: Median (Inter-Quartile Range); unit: μm
Arm/Group | Previous Denosumab
Number analyzed (Participants) | 14
μm | 7.675 [6.680 to 11.880]

11. Secondary Outcome: Bone Histomorphometry: Wall Thickness
Description: Wall thickness is the average thickness of trabecular bone structural units (BSU) and is used to assess the overall balance between resorption and formation.
Time Frame: 25-34 days post-Day 1
Population: All enrolled patients with at least one biopsy evaluable for histomorphometry.
Measure: Median (Inter-Quartile Range); unit: μm
Arm/Group | Previous Denosumab
Number analyzed (Participants) | 14
μm | 40.30 [38.10 to 53.30]

12. Secondary Outcome: Bone Histomorphometry: Eroded Surface/Bone Surface
Description: Eroded surface is expressed as a percentage of total bone surface.
Time Frame: 25-34 days post-Day 1
Population: All enrolled patients with at least one biopsy evaluable for histomorphometry.
Measure: Median (Inter-Quartile Range); unit: percentage of bone surface
Arm/Group | Previous Denosumab
Number analyzed (Participants) | 14
percentage of bone surface | 0.525 [0.300 to 1.110]

13. Secondary Outcome: Bone Histomorphometry: Osteoclast Number - Length Based
Description: Osteoclast number expressed per mm of bone. Osteoclast number was measured using fluorochrome labeling with tetracyclene and tartrate-resistant acid phosphatase stain (TRAP) staining techniques.
Time Frame: 25-34 days post-Day 1
Population: All enrolled patients with at least one biopsy evaluable for histomorphometry.
Measure: Median (Inter-Quartile Range); unit: 1/mm
Arm/Group | Previous Denosumab
Number analyzed (Participants) | 14
1/mm
  Fluorochrome labeling | 0.150 [0.047 to 0.214]
  TRAP staining | 0.122 [0.070 to 0.250]

14. Secondary Outcome: Bone Histomorphometry: Osteoclast Number - Surface Based
Description: Osteoclast number expressed per bone surface area. Osteoclast number was measured using fluorochrome labeling with tetracyclene and tartrate-resistant acid phosphatase stain (TRAP) staining techniques.
Time Frame: 25-34 days post-Day 1
Population: All enrolled patients with at least one biopsy evaluable for histomorphometry.
Measure: Median (Inter-Quartile Range); unit: 1/100 mm
Arm/Group | Previous Denosumab
Number analyzed (Participants) | 14
1/100 mm
  Fluorochrome labeling | 15.0 [14.7 to 21.4]
  TRAP staining | 12.2 [7.0 to 25.0]

15. Secondary Outcome: Bone Histomorphometry: Single-label Surface
Description: Single-label surface is expressed as a percentage of total bone surface. The presence of a single label indicates that mineralization was occurring during only one labeling period.
Time Frame: 25-34 days post-Day 1
Population: All enrolled patients with at least one biopsy evaluable for histomorphometry.
Measure: Median (Inter-Quartile Range); unit: percentage of bone surface
Arm/Group | Previous Denosumab
Number analyzed (Participants) | 14
percentage of bone surface | 2.655 [1.520 to 3.550]

16. Secondary Outcome: Bone Histomorphometry: Double-label Surface
Description: Double-label surface is expressed as a percentage of total bone surface. The presence of double labels indicates that normal bone mineralization was actively occurring over the labeling interval.
Time Frame: 25-34 days post-Day 1
Population: All enrolled patients with at least one biopsy evaluable for histomorphometry.
Measure: Median (Inter-Quartile Range); unit: percentage of bone surface
Arm/Group | Previous Denosumab
Number analyzed (Participants) | 14
percentage of bone surface | 2.895 [1.610 to 4.230]

17. Secondary Outcome: Bone Histomorphometry: Total Mineralizing Surface
Description: Total mineralizing surfaces (MS) include all double and half of single-labeled surfaces. MS is expressed as a percentage of total bone surface.
Time Frame: 25-34 days post-Day 1
Population: All enrolled patients with at least one biopsy evaluable for histomorphometry.
Measure: Median (Inter-Quartile Range); unit: percentage of bone surface
Arm/Group | Previous Denosumab
Number analyzed (Participants) | 14
percentage of bone surface | 4.470 [3.130 to 5.880]

18. Secondary Outcome: Bone Histomorphometry: Mineral Apposition Rate
Description: The mineral apposition rate (MAR) is the avarage rate at which new bone mineral is being added on any actively forming surface. MAR is calculated as the average distance between visible labels, divided by the labeling interval.
Time Frame: 25-34 days post-Day 1
Population: All enrolled patients with at least one biopsy evaluable for histomorphometry.
Measure: Median (Inter-Quartile Range); unit: μm/day
Arm/Group | Previous Denosumab
Number analyzed (Participants) | 14
μm/day | 0.740 [0.630 to 0.890]

19. Secondary Outcome: Bone Histomorphometry: Adjusted Mineral Apposition Rate
Description: The mineral apposition rate (MAR) is the avarage rate at which new bone mineral is being added on any actively forming surface. Adjusted MAR is calculated as: (average distance between visible labels / labeling interval) * (total mineralizing surface/total bone surface).
Time Frame: 25-34 days post-Day 1
Population: All enrolled patients with at least one biopsy evaluable for histomorphometry.
Measure: Median (Inter-Quartile Range); unit: μm/day
Arm/Group | Previous Denosumab
Number analyzed (Participants) | 14
μm/day | 0.750 [0.410 to 1.340]

20. Secondary Outcome: Bone Histomorphometry: Bone Formation Rate - Surface Based
Description: Bone formation rate - surface based (BFR/BS) is the calculated rate at which cancellous bone surface is being replaced annually. BFR/BS is derived from the Mineral Appositional Rate * 365 * (relative mineralizing surface /total bone surface).
Time Frame: 25-34 days post-Day 1
Population: All enrolled patients with at least one biopsy evaluable for histomorphometry.
Measure: Median (Inter-Quartile Range); unit: μm^3 /μm^2 /year
Arm/Group | Previous Denosumab
Number analyzed (Participants) | 14
μm^3 /μm^2 /year | 11.930 [10.560 to 14.860]

21. Secondary Outcome: Bone Histomorphometry: Bone Formation Rate - Volume Based
Description: Bone formation rate - volume based (BFR/BV) is the calculated rate at which cancellous bone volume is being replaced annually. BFR/BV is derived from the Mineral Appositional Rate * 365 * (relative mineralizing surface / total bone volume).
Time Frame: 25-34 days post-Day 1
Population: All enrolled patients with at least one biopsy evaluable for histomorphometry.
Measure: Median (Inter-Quartile Range); unit: percent of bone volume per year
Arm/Group | Previous Denosumab
Number analyzed (Participants) | 14
percent of bone volume per year | 18.780 [12.050 to 27.340]

22. Secondary Outcome: Bone Histomorphometry: Formation Period
Description: The formation period is the duration of an interval when a place on the bone surface is actively forming bone. The formation period is calculated as the wall width (thickness of new bone made in one cycle) divided by the mineral apposition rate.
Time Frame: 25-34 days post-Day 1
Population: All enrolled patients with at least one biopsy evaluable for histomorphometry.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Previous Denosumab
Number analyzed (Participants) | 14
days | 60.7 [32.4 to 88.4]

23. Secondary Outcome: Bone Histomorphometry: Activation Frequency
Description: The average time that it takes for a new remodeling cycle to begin on any point on a cancellous surface is called the activation frequency (Ac.f). Activation frequency is calculated as the bone formation rate / wall width.
Time Frame: 25-34 days post-Day 1
Population: All enrolled patients with at least one biopsy evaluable for histomorphometry.
Measure: Median (Inter-Quartile Range); unit: /year
Arm/Group | Previous Denosumab
Number analyzed (Participants) | 14
/year | 0.261 [0.198 to 0.360]

24. Secondary Outcome: Bone Histomorphometry: Osteoid Volume
Description: Osteoid volume is expressed as a percentage of total bone volume.
Time Frame: 25-34 days post-Day 1
Population: All enrolled patients with at least one biopsy evaluable for histomorphometry.
Measure: Median (Inter-Quartile Range); unit: percentage of total volume
Arm/Group | Previous Denosumab
Number analyzed (Participants) | 14
percentage of total volume | 0.515 [0.120 to 1.360]

25. Secondary Outcome: Bone Histomorphometry: Mineralization Lag Time
Description: The mineralization lag time is the time interval between osteoid secretion and its subsequent mineralization, in days.
Time Frame: 25-34 days post-Day 1
Population: All enrolled patients with at least one biopsy evaluable for histomorphometry.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Previous Denosumab
Number analyzed (Participants) | 14
days | 11.9 [7.6 to 19.9]

26. Secondary Outcome: C-Telopeptide (CTX-1)
Description: C-Telopeptide is a biochemical marker for bone turnover. Blood samples were drawn for assessment of CTX-1 levels on either Day 3 or Day 20, within 24 hours of the last dose of the respective tetracycline cycle.
Time Frame: Day 3 or Day 20
Population: All enrolled patients with at least one evaluable biopsy
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | Previous Denosumab
Number analyzed (Participants) | 15
ng/mL | 0.646 [0.494 to 0.789]

27. Secondary Outcome: Procollagen Type 1 N-terminal Peptide (P1NP)
Description: Procollagen Type 1 N-terminal Peptide is a biochemical marker of bone turnover. Blood samples were drawn for assessment of P1NP levels on either Day 3 or Day 20, within 24 hours of the last dose of the respective tetracycline cycle.
Time Frame: Day 3 or Day 20
Population: All enrolled patients with at least one evaluable biopsy
Measure: Median (Inter-Quartile Range); unit: μg/L
Arm/Group | Previous Denosumab
Number analyzed (Participants) | 15
μg/L | 50.70 [40.80 to 58.90]

ADVERSE EVENTS:
Time Frame: up to 50 days
Description: The table of Other Adverse Events summarizes the most frequent non-serious occurrences of adverse events.
Arm/Group | Previous Denosumab
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 15/15
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Previous Denosumab (N=15)
Dyspepsia (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 1
Post procedural haematoma (Injury, poisoning and procedural complications) | 6
Procedural pain (Injury, poisoning and procedural complications) | 12
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Hypoaesthesia (Nervous system disorders) | 1
Hot flush (Vascular disorders) | 2
Hypertension (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multi-center studies, the investigator agrees not to publish any results before the first multi-center publication.